CLINICAL TRIAL: NCT06055283
Title: Effects of Intradialytic Aerobic Exercise on Peripheral Muscle Function, Functional Status and Motivation in Chronic Kidney Patients: A Randomized Controlled Clinical Trial
Brief Title: Effects of Intradialytic Aerobic Exercise in Chronic Kidney Patients
Acronym: IAECKD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Jéssica Canizelli Gonçalez, doctoral student, University of the State of Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECRC/CKD
Record Dates: First submitted 2023-06-05; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): Aerobic exercise training on moderate intensity.
  Interventions: Other: Aerobic exercise
- Control group (No Intervention): Monitoring.

INTERVENTIONS:
Other: Aerobic exercise — The training group will receive aerobic exercise and the intensities will be controlled considering the percentage of estimated maximum heart rate. The training will be performed with a cycle ergometer with a total of 40 minutes of intradialytic aerobic exercise in the training group. To reduce the effects of intolerance to aerobic exercise, a week of adaptation will be performed, with a frequency of three sessions, in the first two hours of hemodialysis, lasting 40 minutes at maximum heart rate intensity of up to 74% and BORG up to 4 (low intensity). Afterwards, the patients will perform the prediction training for 12 weeks, at the frequency of three training sessions per week in the first two hours of hemodialysis. Each training session will start with a 5-minute warm-up at low intensity, 30 minutes of main training with maximum heart rate intensity 55% to 74% and BORG 5 to 7 (moderate intensity) and will end with a 5-minute cool-down at low intensity.
  Arms: Training group

SUMMARY:
The goal of this clinical trial is to evaluate the effects of intradialytic aerobic exercise on muscle capacity, functionality and motivation of patients with chronic kidney disease undergoing hemodialysis.

The main question it aims to answer are:

• Is intradialytic aerobic exercise at moderate intensity effective in improving peripheral muscle function, functional status and motivation in patients with chronic kidney disease?

DETAILED DESCRIPTION:
The progressive and irreversible advance of chronic kidney disease generates the systemic involvement of the organism and, consequently, the impairment of functionality and quality of life. Hemodialysis therapy is a strategy to increase survival and its long implementation time appears as a space for physiotherapeutic interventions in delaying functional impairment in these individuals. The objective will be to evaluate the effects of intradialytic aerobic exercise on muscle capacity, functionality and motivation of patients with chronic kidney disease undergoing hemodialysis. Patients with chronic kidney disease who undergo hemodialysis at TR São José - Clínica de hemodialysis LTDA (São José/SC) will be evaluated. Patients will be randomized, via a convenience sample, into two groups: intradialytic aerobic exercise group and control group. Interventions will take place within the first two hours of hemodialysis, using a portable cycle ergometer. Intensity will be controlled by heart rate and BORG Perceived Exertion Index. The training, for both groups, will be three times a week, for a period of three months. The aerobic exercise intensity will be moderate, in the percentage of maximum heart rate from 55 to 74% and BORG 4 to 6. A portable cycle ergometer will be used. The evaluations will be in the baseline period, after each complete month and after six months of the end. There will be three days of assessments at the hemodialysis clinic prior to renal replacement therapy and seven days using a home device, following the sequence: baseline blood sample collection, anthropometric assessment, vital signs, BORG, spirometry, mean quadriceps thickness, capacity functional status (six-minute step test), cognitive status (Montreal Cognitive Assessment-BR), quality of life (Kidney Disease And Quality-Of-Life Short Form), sleep quality (Pittsburgh Sleep Quality Index), state motivational (Behavior Regulation Exercise Questionnaire - BREQ3), muscle strength and endurance and daily physical activity. The sample calculation will be performed a posteriori, with Gpower software, based on the variables of the six-minute step test and muscle resistance value. Data will be systematized in the Statistical Package for Social Sciences version 20.0. Initially, descriptive statistics will be performed. To characterize the sample, the following variables will be considered: age, gender, anthropometric data, spirometric parameters, body composition, urea and creatinine clearance, cognitive status. Data distribution will be evaluated using the Shapiro-Wilk test or a non-parametric analogue. To compare the response of the outcome variables between the groups, the ANOVA two-way test of repeated measures, or a non-parametric analogue, will be used. To verify relationships between numeric variables, Pearson's correlation coefficient or non-parametric analogue will be used. The significance level adopted for the statistical treatment will be 5% (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic kidney disease undergoing renal replacement therapy via hemodialysis
* aged 20 to 65 years
* low body mass index at overweight (21 kg/m2 to 29.9 kg/m2)
* regular renal replacement therapy via hemodialysis for 6 months, without acute complications related to the diagnosis and/or comorbidities for the period of 3 months prior to the evaluation and intervention.

Exclusion Criteria:

* patients who do not reach a score equal to or above 20 assessed by the Mini Mental State Examination
* severe heart failure according to the New York Heart Association classification
* musculoskeletal alteration that prevents the correct execution of the assessment activities
* who have participated in other exercise protocols in the last 6 months prior to the present study
* patients who show signs of clinical instability during the hemodialysis procedure or after training for two consecutive sessions will be excluded throughout the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-06-14 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
six minute step test | 12 weeks
  A step 20 centimeters high will be used and the patient will be instructed to go up and down it as many times during the 6 minutes, according to free cadence and will be instructed not to use the upper limbs

SECONDARY OUTCOMES:
muscle strength | 12 weeks
  measured by dynamometry, the records will be in newtons.
Daily life physical activity | 12 weeks
  number of steps for seven days by triaxial accelerometer
Behavior Regulation Questionnaire for Physical Exercise | 12 weeks
  The questionnaire ranges from 0 to 24 for self-regulation indices and 0 to 4 for each type of regulation, namely external, introjected, identified, integrated and intrinsic regulation
index of self-determination and basic psychological needs | 12 weeks
  The score varies from 1 to 5, with 1 being total disagreement and 5 total agreement for variables related to the link between competence and autonomy.
Pittsburg Sleep Quality Index | 12 weeks
  The questionnaire quantifies sleep quality, calculated between seven skills. The final result varies from good sleep quality (0-4), poor sleep quality (5-10) and the presence of sleep disorders (above 10).
Montreal Cognitive Assessment | 12 weeks
  8 cognitive domains (visual-spatial execution, naming, memory, attention, language, abstraction, delayed recall and orientation), with a score from 0 to 30. The cut-off point for renal hemodialysis patients is less than or equal to 24, and the the higher the score, the better the vascular cognitive function
blood sample | 12 weeks
  The analyzes carried out will be regarding the marker of muscle trophism (insulin-like growth factor type 1), pro-inflammatory cytokines (tumor necrosis factor - TNF-alpha) and anti-inflammatory cytokines (interleukin 10 - IL-10).
lower limb resistance | 12 weeks
  Measured by dynamometry, the records will be in tolerated seconds.
Kidney Disease and Quality-of-Life - Short Form | 12 weeks
  eight dimensions, ten items for physical functioning, four items for limitations caused by physical health problems, three items for limitations caused by emotional health problems, two items for social functioning, five items for mental health, two items for pain, four items for vitality, energy and fatigue, five items for perceptions of general health and one item for current health status compared to a year ago, which is computed separately.The degree of commitment is measured using values ranging from zero (highest degree of commitment) to 100 (no commitment). Therefore, the higher the score obtained, the better the quality of life.

IPD SHARING:
Plan to Share IPD: No